CLINICAL TRIAL: NCT06743438
Title: Long-term Safety and Efficacy of Tenofovir Amibufenamide in Patients With HBeAg-positive or HBeAg-negative Chronic Hepatitis B - a Multicenter, Open-label Follow-up Study
Brief Title: Long-term Safety and Efficacy of Tenofovir Amibufenamide in Patients With CHB
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10234-401
Record Dates: First submitted 2024-12-13; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic；HBV infection
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMF treatment group (Experimental)
  Interventions: Drug: Tenofovir Amibufenamide（TMF）

INTERVENTIONS:
Drug: Tenofovir Amibufenamide（TMF） — Once-daily oral dose of 25 mg TMF were maintained in all participants
  Other Names: HS-10234

SUMMARY:
Tenofovir amibufenamide (TMF) is a novel prodrug of tenofovir that has been widely used in mainland China for the treatment of chronic hepatitis B (CHB). The previous registrational study (NCT03903796) has established the non-inferior virologic efficacy of TMF to tenofovir disoproxil fumarate (TDF), while demonstrating higher rates of alanine aminotransferase (ALT) normalization and improved bone and renal safety profiles. This study presented the long-term efficacy and safety of TMF in a phase IV study.

DETAILED DESCRIPTION:
Participants from the Phase III registrational trial of TMF were enrolled and followed for another seven years, starting at week 144 in the Phase III study as the baseline. Once-daily oral dose of 25 mg TMF were maintained in all participants. Clinical assessments were conducted every 24 weeks. The primary efficacy endpoint was the percentage of patients with serum HBV DNA levels below the quantification limit at week (144+) 96.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HBeAg-positive or HBeAg-negative chronic hepatitis B who completed a pivotal Phase III clinical study of HS-10234-301

Exclusion Criteria:

* 1) Completion of HS-10234-301 pivotal Phase III clinical study Interruption of TMF treatment for more than 24 weeks or continuous use of alternative, commercially available hepatitis B antivirals for more than 24 weeks (Participants who have discontinued TMF for more than 24 weeks can only be enrolled in this study after investigator evaluation and confirmation) 2）Evidence of hepatocellular carcinoma (e.g. as evidenced by recent imaging). 3)significant bone disease (e.g. osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochrondroses), or multiple bone fractures.

  4）Currently receiving therapy with immunomodulators (e.g. corticosteroids), investigational agents, nephrotoxic agents, or agents capable of modifying renal excretion.

  5）Known hypersensitivity to study drugs, metabolites, or formulation excipients.

  6) In the investigator's judgment, current alcohol or substance abuse may interfere with the subject's compliance with the study requirements 7）Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation the percentage of Participants with Hepatitis B Virus (HBV) DNA lower than in the central laboratory | week (144+)96
  The primary efficacy endpoint was the proportion of patients with HBV DNA lower than in the central laboratory at week (144+)96.

SECONDARY OUTCOMES:
The proportion of subjects with HBV DNA with lower than in the central laboratory | week(144+)240、week(144+)336
  The proportion of patients with HBV DNA lower than in the central laboratory at week(144+)240、week(144+)336
Proportion of subjects with ALT normalization rate | week (144+)96、week (144+)240、week (144+)336
  The proportion of patients with normal ALT
Proportion of Patients Achieving HBsAg loss，HBsAg conversion | week (144+)96、week (144+)240、week (144+)336
  The denominator of HBsAg loss was the number of HBsAg- positive patients at 144 weeks. The denominator of HBsAg seroconversion was the number of HBsAg positive and anti-HBs negative persons at 144 weeks.
Incidence of resistance mutation | week (144+)96、week (144+)240、week (144+)336
  Resistance detection when a virological breakthrough occurs
Progression of liver disease associated with HBV infection | week (144+)96、week (144+)240、week (144+)336
  The proportion of patients with new HCC, Decompensated liver cirrhosis, death related to Hepatitis B
Proportion of Patients Achieving HBeAg loss，HBeAg conversion ratio | week (144+)96、week (144+)240、week (144+)336
  The denominator of HBeAg loss was the number of HBeAg- positive patients at 144 weeks. The proportion of HBeAg seroconversion was the number of HBeAg positive and anti-HBs negative persons at 144 weeks.
Percent Change from Baseline in Hip and spine Bone Mineral Density (BMD) | week (144+)96、week (144+)240、week (144+)336
  measured by dual energy x-ray absorptiometry(DXA)
Change from Baseline in Serum Creatinine | week (144+)96、week (144+)240、week (144+)336
Change in HBV DNA from baseline | week (144+)96、week (144+)240、week (144+)336

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, M.M, Principal Investigator — Nanfang Hospital, Southern Medical University; Junqi Niu, MD, Principal Investigator — The First Hospital of Jilin University; Guicheng Wu, MD, Principal Investigator — Chongqing University Affiliated Three Gorges Hospital; Peng Hu, MD, Principal Investigator — The second affiliated hospital of chongqiong medical university; Lvfeng Yao, Principal Investigator — Mengchao Hepatopiliary Hospital of Fujian Medical University; Wenhong Zhang, MD, Principal Investigator — Huashan Hospital; Minghua Su, MM, Principal Investigator — First Affiliated Hospital of Guangxi Medical University; Xiaoqing Fu, MM, Principal Investigator — Hangzhou Xixi hospital; Caiyan Zhao, MD, Principal Investigator — Third hospital of Hebei Medical University; Jia Shang, Principal Investigator — Henan Provincial People's Hospital; Xiaorong Mao, MD, Principal Investigator — LanZhou University; Shufang Yuan, MD, Principal Investigator — LiuZhou People's Hospital; Jie Li, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Qing Xie, MD, Principal Investigator — Ruijin Hospital; Qin Zhang, MD, Principal Investigator — Tongren Hospital,Shanghai Jiao Tong University School of Medicine; Desheng Xie, MM, Principal Investigator — Shanghai Fifth People's Hospital; Liang Chen, MM, Principal Investigator — Shanghai Public Health Clinical Center; Yao Xie, MD, Principal Investigator — Beijing Ditan Hospital; Jidong Jia, MD, Principal Investigator — Beijing Friendship Hospital; Enqiang Chen, MD, Principal Investigator — West China Hospital; Xingxiang Yang, MM, Principal Investigator — Sichuan Academy of Medical Sciences; Fengmei Wang, MD, Principal Investigator — Tianjin Third Central Hospital; MingQin Lu, MM, Principal Investigator — The First Hospital of Wenzhou Medical University; Lihua Sun, MD, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Daokun Yang, MM, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Xuebing Yan, MD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Huazhong Chen, MM, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University; Min Zhang, MD, Principal Investigator — Central South University; Yan Huang, MD, Principal Investigator — Xiangya Hospital of Central South University; Yawen Luo, MM, Principal Investigator — Zunyi Medical College; Lihua Zhong, MM, Principal Investigator — The Fourth Affiliated Hospital of Harbin Medical University; Min Xie, Principal Investigator — Guangzhou Eighth People's Hospital; Jun Li, MD, Principal Investigator — Jiangsu Provincial People's Hospital (The First Affiliated Hospital of Nanjing Medical University)
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided